CLINICAL TRIAL: NCT00603772
Title: Clinical Evaluation of the Photoallergy Potential of Atralin Gel (Tretinoin Gel 0.05%)
Brief Title: Clinical Evaluation of the Photoallergy Potential of Atralin Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coria Laboratories, Ltd. (Industry)
Responsible Party: D. Innes Cargill, PhD, Coria Laboratories, Ltd.
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 029-066-09-002
Record Dates: First submitted 2008-01-08; First posted 2008-01-29 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-02

CONDITIONS: Healthy
Keywords: Tretinoin; exposure to UV light; phototoxicity; Safety when exposed to sunlight
MeSH Terms: conditions — Dermatitis, Phototoxic | interventions — Tretinoin; Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Safety when exposed to sunlight
  Interventions: Drug: Atralin (tretinoin) gel, 0.05%

INTERVENTIONS:
Drug: Atralin (tretinoin) gel, 0.05% — Assess photoallergic reactions for tretinoin 0.05% and vehicle, measured as skin reactions following induction and challenge.

SUMMARY:
To assess the potential of tretinoin gel 0.05% and its vehicle to produce photoallergic reactions, measured as skin reactions following induction and challenge.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy volunteers
* 18 years of age and older

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
UV Induced skin irritation | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Stanfield, MS, Principal Investigator — Suncare Research Laboratories
Locations (1):
- Suncare Research Laboratories, Winston-Salem, North Carolina, United States